CLINICAL TRIAL: NCT01643733
Title: Confirmation of Clinical Effectiveness and Safety of Use of Transonics in Determining Success of Intervention in Dialysis Fistulae
Brief Title: Study on Fistuloplasty Using Flow Measurement Guidance
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough recruitment
Sponsor: Richard Lindsay (Other)
Responsible Party: Sponsor-Investigator, Richard Lindsay, MD, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-133-SDR
Record Dates: First submitted 2012-07-10; First posted 2012-07-18 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: End Stage Renal Failure on Dialysis; Renal Failure
Keywords: Angioplasty
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transonics Arm (Experimental): Intervention will be guided by flow through the fistula as guided by Transonics flow measurements
  Interventions: Device: Using Flow measurements to guide fistula angioplasty (Transonics)
- Control arm (No Intervention): Patient will undergo normal fistula intervention guided only by angiographic assessment

INTERVENTIONS:
Device: Using Flow measurements to guide fistula angioplasty (Transonics) — Transonics flow measurements in the fistula would be used to guide the fistula intervention
  Arms: Transonics Arm

SUMMARY:
Hypothesis: The primary objective of this study is to assess whether using a flow measurement device, in this case the Transonics flow device, as an end-point to interventional treatment of diseased dialysis fistulae can help increase immediate treatment success in terms of quality of dialysis immediately following the treatment and increasing time to reintervention.

DETAILED DESCRIPTION:
This is a prospective randomized study. All intervention will be carried out by experienced radiologists in the two study centres.

At least fifty (50) consecutive subjects meeting the eligibility criteria, scheduled for angiographic assessment (with a view to PTA if necessary), will be invited to participate in the study. Subjects who consent will undergo their procedure, which will be performed by a qualified interventional radiology doctor (IRD). Patients will be randomly allocated to each group. All previous Transonics measurements will be available to the treating IRD. A target flow rate will be pre-decided in all patients in consultation with the nephrology service.

* All patients will undergo a fistulogram, a routine interventional Xray exam where radiocontrast media (RCM) is injected under X ray control to identify narrowings within the vessels. Significant lesions will be identified based on this exam. If a lesion is believed to be significant, the patient will be assigned to either arm of the study. The details of the disease present will be recorded as location and percentage stenosis.
* In the control arm, an initial Transonic measurement pre-treatment will be performed. The interventionalist will select the most significant lesion based on angiographic appearances and treat this lesion, which may require use of multiple balloons for the same lesion. At this point a Transonics measurement will be taken - Measurement A. The results will not be revealed to the interventionalist, who will proceed with the procedure as per their standard practice. A Transonics measurement will be taken after treatment of each of the significant lesions identified at the start of the exam. A post-procedural Transonics measurement (Measurement X) will also be taken, again the interventionalist will blinded as to this result. The appearances on completion angiography will be recorded as percentage stenosis remaining.
* In the Transonics arm, a pre-treatment Transonic measurement will be done. The lesions will be treated. Once Measurement A is obtained, the interventionalist will only be informed if the target value has been reached or not, they will not be told the actual value. This will be repeated for the treatment of each subsequent lesion, with the interventionalist being informed if the target had been reached, whilst being blinded as to the Transonics result, until the target has been achieved. The interventionalist will not pursue further treatment, regardless of the Transonics measurement, if he deems it would pose a greater risk of complication to the patient, than his/her standard practice. The appearances on completion angiography will be recorded as percentage stenosis remaining.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female subjects, between the ages of 18 and 80 at the time of enrollment.
* Subjects referred to us from the Dialysis units located in the study centres for clinically indicated fistulogram and fistula treatment.
* Written informed consent to participate in the study.
* Ability to comply with the requirements of the study procedures

Exclusion Criteria:

* Significant coagulopathy that cannot be adequately corrected.
* Subjects who participated in an active stage of any drug, intervention or treatment trial within 30 days of enrollment.
* Subjects with preexisting conditions, which, in the opinion of the investigator, interfere with the conduct of the study. Patients will only be excluded on this basis following discussion with another interventional radiologist and the referring nephrologist.
* Subjects who are uncooperative or cannot follow instructions.
* Mental state that may preclude completion of the study procedure or ability to obtain informed consent.
* Pregnant or nursing female subjects.
* Patients whose fistulae have never become functional.
* Patients with PTFE grafts/non-native fistulae
* Patients who have had previous stenting of fistulae

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-10; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Time to reintervention | 6 months
  Time between intervention and the need for repeat intervention (based on standard dialysis screening systems).

SECONDARY OUTCOMES:
Effect of treatment on rate of change in Transonics flow measurements | Baseline, 2 weeks, one, two three and 6 months
  Analysis of Transonics flow measurements obtained post intervention during the follow-up of six months
Change in dialysis efficiency post treatment | One month, 2, 3 and six months
  Comparison of Dialysis efficiency scores pre and post treatment
Significance of stenoses as detected by Transonics, compared with angiography | 1 day, ie.will be asessed immediately following intial intervention only.
  Assessment of extent to which using flow measurements can improve ability to detect hemodynamically significant stenoses.
Nature of Procedure using Transonics versus Angiographic assessment | Six months
  Comparison of procedures carried out between the group where Transonics flow measurements are used to guide intervention, versus the group where angiographic assessment is used.

CONTACTS AND LOCATIONS:
Overall Officials: David Valenti, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Louis Boucher, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (2):
- Canada (2):
  - Royal Victoria Hospital, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec